CLINICAL TRIAL: NCT06742047
Title: Implementing a Professional Development Programme (ProDeveloP): an Introduction for Newly Graduated Nurses
Brief Title: A Professional Development Programme (ProDeveloP) for Newly Graduated Nurses
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Mälardalen University (Other)
Collaborators: Region Västmanland (Other); AFA Insurance (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 220065
Record Dates: First submitted 2024-12-18; First posted 2024-12-19 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-12

CONDITIONS: Professional Fulfillment; Professional Identity Formation; Professional Quality of Life; Support Program; Development; Nurse Role
Keywords: Introduction programme; Newly graduated nurses; Professional development; Role clarity; Task mastery; Stress; Recovery; Reflection; Social acceptance; Transition support; Dialogue group; Registered nurse; Focus group; Intervention; Interview; Intensive measures
MeSH Terms: conditions — Social Identification

STUDY DESIGN:
Intervention Model Description: Two cohorts of NGNs received the ProDevelop intervention in 2023 and 2024. A control group in 2022 did not receive the intervention but the previous introduction programme.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Participating in the Professional development program (ProDeveloP) (Experimental): The group received the intervention of the Professional Development Programme (ProDeveloP). The planning of the ProDeveloP has been done in close collaboration with stakeholders within the hospital setting where the programme will be implemented. The programme includes face-to-face approaches from peer learning and e-learning modalities.
  Interventions: Behavioral: Professional development programme
- Control group prior the intervention in 2022 (No Intervention): The group did not receive the intervention

INTERVENTIONS:
Behavioral: Professional development programme — The professional development programme include dialogue groups facilitated by registered nurses (RN) who are expert and experienced supervisors that received a three day training before conducting the groups. Then including education days with joint lectures and simulations with experts in the field with experience. The programme provides NGNs with regular opportunities for reflection for learning from experiences of care to enhance personal and professional growth.
  Arms: Participating in the Professional development program (ProDeveloP)

SUMMARY:
This clinical study aims to implement and evaluate a professional development programme (ProDeveloP) designed to facilitate the transition of newly graduated nurses (NGNs) into their new roles. NGNs face several challenges in the work environment and in developing their professional competencies. The aim is to support NGNs in a county hospital in central Sweden to facilitate their professional development. Data will be collected during the NGNs' first year through intensive longitudinal measures, including weekly and quarterly questionnaires. This will be combined with individual interviews and focus groups with NGNs, dialogue facilitators and managers.

DETAILED DESCRIPTION:
The primary outcomes will be role clarity, task mastery, social acceptance, recovery and stress. The researchers will compare the results of the primary outcomes with those of a control group measure. Secondary outcomes will be experience of the intervention, transition support, job satisfaction and intention to leave.

Informed consent was signed prior to participation in the study. The ethical application has been approved by the Ethics Authority IS, diary number 2022-05682-0.

ELIGIBILITY:
Inclusion criteria:

* Registered nurses in Sweden employed as Newly Graduated Nurses (NGNs) in a county in central Sweden participating in the ProDeveloP, the intervention group.
* Registered nurses in Sweden employed as Newly Graduated Nurses (NGNs) in a county in central Sweden, NGNs participating in the introduction programme prior to the study, not participating in the ProDeveloP, the control group.
* Experienced registered nurses as facilitators for the dialogue groups for the NGNs in the intervention.
* Managers at the county hospital for the NGNs participating in the intervention.

Exclusion criteria:

• Managers without NGNs participated in the intervention.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2023-02-06 (Actual); Primary Completion 2024-09-17 (Actual); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Role Clarity | The measurement was carried out thirteen times, every week during the first time participation in the ProDeveloP intervention. The control group was measured at the thirteenth week after the start of the introduction programme.
  The professional development process in terms of gaining clarity about the responsibilities content and boundaries of the role. Validated questions from the Questionnaire for Psychological and Social Factors at Work (QPS Nordic). 5-point Likert scale.
  During the last week, how did you feel about:
  Having clearly defined goals? You know what your responsibilities are? You know exactly what is required of you at work?
Recovery | The measurement was carried out thirteen times, every week during the first time participation in the ProDeveloP intervention and then at months 4, 8 and 12 after the start. The control group was measured at the thirteenth week.
  Thirteen weekly and three monthly measures. 5-point Likert scale. Experience of rest, In the past week I was able to relax? and at home including leisure activities, In the past week, I was able to do activities that give me energy? Validated questions on sleep from the Karolinska Sleep Questionnaire on sleep. How did you sleep last night? During the past week, did you find it difficult to let go of thoughts about work in your free time? Validated questions from QPS Nordic, How did you feel about the workload during the last week?
  For the three monthly measurements. 5-point Likert scale. Questions from the Balancing Work with Recovery scale, In the last month, how often have you felt rested and recovered after a weekend or two-day holiday? Do the demands of your work have a negative impact on your personal life?
Task Mastery | The measurement was carried out thirteen times, every week during the first time participation in the ProDeveloP intervention. The control group was measured at the thirteenth week after the start of the introduction programme.
  The development of skills and experience to complete their work tasks and handle the more complex tasks. Validated questions from the Needs Satisfaction and Frustration Scale (NSFS). 5-point lickert scale. During the last week: I have felt that I have been able to fulfill even the most demanding tasks? I have felt that I have been good at doing my job?
Social acceptance | The measurement was carried out thirteen times, every week during the first time participation in the ProDeveloP intervention. The control group was measured at the thirteenth week after the start of the introduction programme.
  Being integrated into the work group and belonging at work with questions from the validated Needs Satisfaction and Frustration Scale (NSFS). 5-point lickert scale. During the last week: I have felt that the people I work with have really cared about me? I have felt included in the work group?
Stress | The measurement was carried out thirteen times, every week during the first time participation in the ProDeveloP intervention and then at months 4, 8 and 12 after the start. The control group was measured at the thirteenth week.
  Stress levels from questions from the validated Stress and Energy Questionnaire (SEQ). 5-point lickert scale. During the last week when you have been working, how often have you felt: Tense? Stressed? Pressured?

SECONDARY OUTCOMES:
Job satiscation | Measured during months 4, 8 and 12 of participating in the intervention.
  Satisfaction of the professional work. 5-point lickert scale. Questions from the validated Job Satisfaction scale. How often do you feel about your work in the following ways : I feel happy at work? I feel satisfied with the work I have? I feel satisfaction with my work?
Intentions to leave | Measured during months 4, 8 and 12 of participating in the intervention.
  Intentions to leave the workplace or profession. 5-point lickert scale. Questions from the validated Organizational Commitment on Job Turnover Intention scale. Please respond to the following statements about changing jobs: I often think about leaving my current place of work?As soon as it is possible, I will leave my current place of work? I am actively looking for a job outside my current workplace? Please comment on the following statements about changing profession: I often think about changing profession? I actively look for work outside this profession? I would like to leave this profession as soon as possible?

CONTACTS AND LOCATIONS:
Overall Officials: Margareta Asp, Professor, Principal Investigator — Mälardalens University
Locations (1):
- Mälardalens University, Västerås, Sweden

IPD SHARING:
Plan to Share IPD: No
The ethical approval do not allow to share IPD outside the research group.

REFERENCES:
- [Derived] Hoglander J, Lindblom M, Sodersved Kallestedt ML, Letterstal A, Asp M, Widarsson M. Implementing a Professional Development Programme (ProDeveloP) for Newly Graduated Nurses: A Study Protocol. Nurs Rep. 2025 Jul 2;15(7):243. doi: 10.3390/nursrep15070243. PMID 40710938